CLINICAL TRIAL: NCT00090311
Title: A 3-wk, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Phase 3b Study of the Efficacy & Safety of Quetiapine Fumarate (SEROQUEL™) Immediate-release Tablets in the Treatment of Children & Adolescents With Bipolar I Mania (Abbreviated)
Brief Title: Quetiapine Fumarate (SEROQUEL) Compared to Placebo in the Treatment of Children & Adolescents With Bipolar I Mania
Acronym: ANCHOR 149
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1441C00149
Record Dates: First submitted 2004-08-25; First posted 2004-08-30 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Mania
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: quetiapine fumarate

SUMMARY:
The purpose of this study is to demonstrate efficacy and safety of quetiapine fumarate (SEROQUEL) compared with placebo in the treatment of children and adolescent patients with Bipolar I mania.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to provide written assent and the parents or legal guardian of the patient is able to provide written informed consent before beginning and study related procedures
* Patient has a documented clinical diagnosis of Bipolar I mania
* Patient's parent or legal guardian will be able to accompany the patient at each scheduled study visit

Exclusion Criteria:

* Patients (female) must not be pregnant or lactating
* Patients with a known intolerance or lack of response to previous treatment with quetiapine
* Patients who have previously participated in this study

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2004-07; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Compare efficacy of Quetiapine with placebo in the treatment of bipolar I mania as assessed by the YMRS total score, change from baseline to Day 21

SECONDARY OUTCOMES:
Compare the effect of Quetiapine with placebo in change from baseline to Day 21 percentage of patients with response, defined as a ≤ 12, evaluate safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (32):
- United States (32):
  - Research Site, Scottsdale, Arizona
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Denver, Colorado
  - Research Site, Alamonte, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, New Orleans, Louisiana
  - Research Site, Saint Charles, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Clementon, New Jersey
  - Research Site, Piscataway, New Jersey
  - Research Site, Rochester, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Lyndhurst, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Madison, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Kirkland, Washington
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Pathak S, Findling RL, Earley WR, Acevedo LD, Stankowski J, Delbello MP. Efficacy and safety of quetiapine in children and adolescents with mania associated with bipolar I disorder: a 3-week, double-blind, placebo-controlled trial. J Clin Psychiatry. 2013 Jan;74(1):e100-9. doi: 10.4088/JCP.11m07424. PMID 23419231